CLINICAL TRIAL: NCT01107886
Title: A Multicentre, Randomised, Double-Blind, Placebo-Controlled Phase IV Trial to Evaluate the Effect of Saxagliptin on the Incidence of Cardiovascular Death, Myocardial Infarction or Ischaemic Stroke in Patients With Type 2 Diabetes
Brief Title: Does Saxagliptin Reduce the Risk of Cardiovascular Events When Used Alone or Added to Other Diabetes Medications
Acronym: SAVOR- TIMI 53
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1680C00003; EudraCT No 2009-017358-10
Record Dates: First submitted 2010-03-25; First posted 2010-04-21 (Estimated); Results first posted 2014-06-13 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2014-07

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Risk of cardiovascular disease and death in patients with type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — saxagliptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Saxagliptin (Experimental)
  Interventions: Drug: Saxagliptin
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Saxagliptin — 5 mg or 2.5 mg once daily
  Other Names: Onglyza
  Arms: Saxagliptin
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether saxagliptin can reduce the risk of cardiovascular events when used alone or added to other diabetes medications

DETAILED DESCRIPTION:
A Multicentre, Randomised, Double-Blind, Placebo-Controlled Phase IV Trial to Evaluate the Effect of Saxagliptin on the Incidence of Cardiovascular Death, Myocardial Infarction or Ischaemic Stroke in Patients with Type 2 Diabetes

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes mellitus
* HbA1c ≥6.5%. (based on the last measured and documented laboratory measurement within 6 months)
* High risk for CV events -Established cardiovascular disease and/or multiple risk factors

Exclusion Criteria:

* Current or previous (within 6 months) treatment with DPP4 inhibitors and/or GLP-1 mimetics
* Acute vascular event <2months prior to randomisation

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18206 (Actual)
Dates: Start 2010-05; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Braunwald, Study Chair — TIMI; Itamar Raz, Principal Investigator — Hadassah Medical Organization; Deepak Bhatt, Principal Investigator — TIMI
Locations (536):
- United States (202):
  - Research Site, Birmingham, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Tempe, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Alhambra, California
  - Research Site, Anaheim, California
  - Research Site, Bakersfield, California
  - Research Site, Burlingame, California
  - Research Site, Duarte, California
  - Research Site, Huntington Park, California
  - Research Site, La Mesa, California
  - Research Site, Lomita, California
  - Research Site, Los Angeles, California
  - Research Site, Oceanside, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, San Ramon, California
  - Research Site, Torrance, California
  - Research Site, Ventura, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, Denver, Colorado
  - Research Site, Longmont, Colorado
  - Research Site, Bridgeport, Connecticut
  - Research Site, Bristol, Connecticut
  - Research Site, Southington, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Coral Springs, Florida
  - Research Site, Daytona Beach, Florida
  - Research Site, Deerfield Beach, Florida
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Green Cove Springs, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Hudson, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Leesburg, Florida
  - Research Site, Miami, Florida
  - Research Site, Naples, Florida
  - Research Site, Oakland Park, Florida
  - Research Site, Ocala, Florida
  - Research Site, Palm Beach Gardens, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Plant City, Florida
  - Research Site, Sarasota, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Tampa, Florida
  - Research Site, Trinity, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Weston, Florida
  - Research Site, Winter Haven, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Conyers, Georgia
  - Research Site, Cumming, Georgia
  - Research Site, Honolulu, Hawaii
  - Research Site, Hayden Lake, Idaho
  - Research Site, Pocatello, Idaho
  - Research Site, Belleville, Illinois
  - Research Site, Chicago, Illinois
  - Research Site, Niles, Illinois
  - Research Site, Avon, Indiana
  - Research Site, Evansville, Indiana
  - Research Site, Fishers, Indiana
  - Research Site, Fort Wayne, Indiana
  - Research Site, Franklin, Indiana
  - Research Site, Greenfield, Indiana
  - Research Site, Valparaiso, Indiana
  - Research Site, Council Bluffs, Iowa
  - Research Site, Newton, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Evansville, Kentucky
  - Research Site, Kenner, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Slidell, Louisiana
  - Research Site, Auburn, Maine
  - Research Site, Bangor, Maine
  - Research Site, Portland, Maine
  - Research Site, Baltimore, Maryland
  - Research Site, Towson, Maryland
  - Research Site, Ayer, Massachusetts
  - Research Site, Boston, Massachusetts
  - Research Site, Haverhill, Massachusetts
  - Research Site, Natick, Massachusetts
  - Research Site, North Dartmouth, Massachusetts
  - Research Site, Alpena, Michigan
  - Research Site, Cadillac, Michigan
  - Research Site, Kalamazoo, Michigan
  - Research Site, Petosky, Michigan
  - Research Site, Pontiac, Michigan
  - Research Site, Rochester, Michigan
  - Research Site, Waterford, Michigan
  - Research Site, Ypsilanti, Michigan
  - Research Site, Baxter, Minnesota
  - Research Site, Chaska, Minnesota
  - Research Site, Duluth, Minnesota
  - Research Site, Eagan, Minnesota
  - Research Site, Minneapolis, Minnesota
  - Research Site, Robbinsdale, Minnesota
  - Research Site, Kansas City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Billings, Montana
  - Research Site, Bellevue, Nebraska
  - Research Site, Fremont, Nebraska
  - Research Site, Grand Island, Nebraska
  - Research Site, Omaha, Nebraska
  - Research Site, Henderson, Nevada
  - Research Site, Las Vegas, Nevada
  - Research Site, Reno, Nevada
  - Research Site, Elizabeth, New Jersey
  - Research Site, Elmer, New Jersey
  - Research Site, Voorhees Township, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Binghamton, New York
  - Research Site, Buffalo, New York
  - Research Site, Cortlandt Manor, New York
  - Research Site, Endwell, New York
  - Research Site, New Hyde Park, New York
  - Research Site, Northport, New York
  - Research Site, Saratoga Springs, New York
  - Research Site, Syracuse, New York
  - Research Site, The Bronx, New York
  - Research Site, Westfield, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Hickory, North Carolina
  - Research Site, Monroe, North Carolina
  - Research Site, Morganton, North Carolina
  - Research Site, Rocky Mount, North Carolina
  - Research Site, Smithfield, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Grand Forks, North Dakota
  - Research Site, Beachwood, Ohio
  - Research Site, Cadiz, Ohio
  - Research Site, Canal Fulton, Ohio
  - Research Site, Canton, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Delaware, Ohio
  - Research Site, Elyria, Ohio
  - Research Site, Kettering, Ohio
  - Research Site, Lorain, Ohio
  - Research Site, Middleburg Hights, Ohio
  - Research Site, Sandusky, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Tulsa, Oklahoma
  - Research Site, Portland, Oregon
  - Research Site, Altoona, Pennsylvania
  - Research Site, Bethlehem, Pennsylvania
  - Research Site, Clymer, Pennsylvania
  - Research Site, Doylestown, Pennsylvania
  - Research Site, Hermitage, Pennsylvania
  - Research Site, Indiana, Pennsylvania
  - Research Site, Jersey Shore, Pennsylvania
  - Research Site, Johnstown, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Sayre, Pennsylvania
  - Research Site, Tyrone, Pennsylvania
  - Research Site, Providence, Rhode Island
  - Research Site, Charleston, South Carolina
  - Research Site, Columbia, South Carolina
  - Research Site, Greer, South Carolina
  - Research Site, Spartenburg, South Carolina
  - Research Site, Rapid City, South Dakota
  - Research Site, Bristol, Tennessee
  - Research Site, Jackson, Tennessee
  - Research Site, Memphis, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Amarillo, Texas
  - Research Site, Arlington, Texas
  - Research Site, Austin, Texas
  - Research Site, Colleyville, Texas
  - Research Site, Dallas, Texas
  - Research Site, Edinburg, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Georgetown, Texas
  - Research Site, Grapevine, Texas
  - Research Site, Houston, Texas
  - Research Site, Irving, Texas
  - Research Site, Katy, Texas
  - Research Site, McAllen, Texas
  - Research Site, Midland, Texas
  - Research Site, Mission, Texas
  - Research Site, Odessa, Texas
  - Research Site, Plano, Texas
  - Research Site, Richardson, Texas
  - Research Site, San Antonio, Texas
  - Research Site, San Marcos, Texas
  - Research Site, Southlake, Texas
  - Research Site, Tomball, Texas
  - Research Site, Victoria, Texas
  - Research Site, Burke, Virginia
  - Research Site, Manassas, Virginia
  - Research Site, Midlothian, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Burien, Washington
  - Research Site, Federal Way, Washington
  - Research Site, Tacoma, Washington
  - Research Site, Wenatchee, Washington
  - Research Site, Milwaukee, Wisconsin
- Argentina (16):
  - Research Site, Buenos Aires
  - Research Site, Ciudad Autonom de Buenos Aires
  - Research Site, CiudadAutonoma de Buenos Aires
  - Research Site, Corrientes
  - Research Site, Córdoba
  - Research Site, La Plata
  - Research Site, Lanus Buenos Aires
  - Research Site, Mar del Plata
  - Research Site, Mendoza
  - Research Site, Morón
  - Research Site, Ramos Mejía
  - Research Site, Rosario
  - Research Site, Rosario Santa Fe
  - Research Site, Santa Fe
  - Research Site, Sarandi Buenos Aires
  - Research Site, Villa Ballester
- Australia (11):
  - Research Site, Ashford
  - Research Site, Fitzroy
  - Research Site, Frankston
  - Research Site, Garran
  - Research Site, Geelong
  - Research Site, Launceston
  - Research Site, Maroubra
  - Research Site, Milton
  - Research Site, Sherwood
  - Research Site, Southport
  - Research Site, Windsor
- Brazil (10):
  - Research Site, Belém
  - Research Site, Brasília
  - Research Site, Campinas
  - Research Site, Curitiba
  - Research Site, Goiânia
  - Research Site, Marília
  - Research Site, Porto Alegre
  - Research Site, Recife
  - Research Site, Rio de Janeiro
  - Research Site, São Paulo
- Canada (34):
  - Research Site, Calgary, Alberta
  - Research Site, Red Deer, Alberta
  - Research Site, Spruce Grove, Alberta
  - Research Site, New Westminster, British Columbia
  - Research Site, Surrey, British Columbia
  - Research Site, Victoria, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Halifax, Nova Scotia
  - Research Site, Brampton, Ontario
  - Research Site, Courtice, Ontario
  - Research Site, Greater Sudbury, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Kingston, Ontario
  - Research Site, Kitchener, Ontario
  - Research Site, London, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, Oshawa, Ontario
  - Research Site, Scarborough Village, Ontario
  - Research Site, Smiths Falls, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Brossard, Quebec
  - Research Site, Chicoutimi, Quebec
  - Research Site, Greenfield Park, Quebec
  - Research Site, Laval, Quebec
  - Research Site, Longueuil, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Saint-Charles-Borromée, Quebec
  - Research Site, Saint-Lambert, Quebec
  - Research Site, Sherbrooke, Quebec
  - Research Site, Regina, Saskatchewan
  - Research Site, Saskatoon, Saskatchewan
- Chile (2):
  - Research Site, Santiago
  - Research Site, Temuco
- China (8):
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Guangzhou
  - Research Site, Hong Kong
  - Research Site, Nanjing
  - Research Site, Shanghai
  - Research Site, Suzhou
  - Research Site, Tianjin
- Czechia (26):
  - Research Site, Beroun
  - Research Site, Blansko
  - Research Site, Brno
  - Research Site, Břeclav
  - Research Site, Cheb
  - Research Site, Chrudim III
  - Research Site, Čáslav
  - Research Site, Havířov
  - Research Site, Hodonín
  - Research Site, Hořovice
  - Research Site, Hradec Králové
  - Research Site, Jablonec nad Nisou
  - Research Site, Kroměříž
  - Research Site, Olomouc-Lazce
  - Research Site, Ostrava
  - Research Site, Ostrava - Belsky Les
  - Research Site, Ostrava-Kunčice
  - Research Site, Ostrava-Vitkovice
  - Research Site, Pardubice
  - Research Site, Pilsen
  - Research Site, Prague
  - Research Site, Přelouč
  - Research Site, Slaný
  - Research Site, Uherské Hradiště
  - Research Site, Valaske Klobouky
  - Research Site, Zlín
- France (10):
  - Research Site, Amiens
  - Research Site, Bron
  - Research Site, Colmar
  - Research Site, Corbeil-Essonnes
  - Research Site, Nantes
  - Research Site, Paris
  - Research Site, Pessac
  - Research Site, Poitiers
  - Research Site, Reims
  - Research Site, Toulouse
- Germany (19):
  - Research Site, Aschaffenburg
  - Research Site, Bad Nauheim
  - Research Site, Bad Oeynhausen
  - Research Site, Berlin
  - Research Site, Deggingen
  - Research Site, Dippoldiswalde
  - Research Site, Dortmund
  - Research Site, Dresden
  - Research Site, Eschweiler
  - Research Site, Giessen
  - Research Site, Goch
  - Research Site, Güglingen
  - Research Site, Hamburg
  - Research Site, Hohenmölsen
  - Research Site, Kassel
  - Research Site, Leipzig
  - Research Site, Mayen
  - Research Site, Rehlingen-Siersburg
  - Research Site, Rotenburg (Wümme)
- Hong Kong (2):
  - Research Site, Hong Kong, Shatin
  - Research Site, Hong Kong
- Hungary (15):
  - Research Site, Balatonfüred
  - Research Site, Békéscsaba
  - Research Site, Budapest
  - Research Site, Cegléd
  - Research Site, Csongrád
  - Research Site, Eger
  - Research Site, Gyöngyös
  - Research Site, Győr
  - Research Site, Gyula
  - Research Site, Miskolc
  - Research Site, Nagykanizsa
  - Research Site, Pécs
  - Research Site, Siófok
  - Research Site, Szolnok
  - Research Site, Veszprém
- India (13):
  - Research Site, Ahmedabad
  - Research Site, Bangalore
  - Research Site, Bengaluru
  - Research Site, Ernakulam District
  - Research Site, Hyderabad
  - Research Site, Indore
  - Research Site, Jaipur
  - Research Site, Mumbai
  - Research Site, Mysore
  - Research Site, Nagpur
  - Research Site, New Delhi
  - Research Site, Pune
  - Research Site, Vadodara
- Israel (14):
  - Research Site, Ashkelon
  - Research Site, Beersheba
  - Research Site, Dimona
  - Research Site, Giv‘atayim
  - Research Site, Haifa
  - Research Site, Holon
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Nahariya
  - Research Site, Petah Tikva
  - Research Site, Rehovot
  - Research Site, Safed
  - Research Site, Tel Aviv
  - Research Site, Ẕerifin
- Italy (20):
  - Research Site, Bergamo
  - Research Site, Catania
  - Research Site, Florence
  - Research Site, Mercato San Severino
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Negrar - VR
  - Research Site, Padua
  - Research Site, Parma
  - Research Site, Pavia
  - Research Site, Pozzuoli
  - Research Site, Prato
  - Research Site, Ravenna
  - Research Site, Roma
  - Research Site, Rozzano
  - Research Site, S Maria Capua Vetere
  - Research Site, San Giovanni Rotondo
  - Research Site, Sessa Aurunca
  - Research Site, Taormina
  - Research Site, Terni
- Mexico (13):
  - Research Site, Aguascalientes
  - Research Site, Culiacán
  - Research Site, Durango
  - Research Site, Guadalajara
  - Research Site, México
  - Research Site, Monclova
  - Research Site, Monterrey
  - Research Site, Nuevo León
  - Research Site, Oaxaca City
  - Research Site, Querétaro
  - Research Site, San Luis Potosí City
  - Research Site, Tijuana
  - Research Site, Xalapa
- Netherlands (22):
  - Research Site, Almelo
  - Research Site, Amersfoort
  - Research Site, Amsterdam
  - Research Site, Apeldoorn
  - Research Site, Arnhem
  - Research Site, Breda
  - Research Site, Delft
  - Research Site, Eindhoven
  - Research Site, Goes
  - Research Site, Gouda
  - Research Site, Groningen
  - Research Site, Hardenberg
  - Research Site, Hoogeveen
  - Research Site, Hoorn
  - Research Site, Leiderdorp
  - Research Site, Nijmegen
  - Research Site, Rotterdam
  - Research Site, Sneek
  - Research Site, Utrecht
  - Research Site, Velp
  - Research Site, Waalwijk
  - Research Site, Zoetermeer
- Peru (3):
  - Research Site, Callao
  - Research Site, Lima
  - Research Site, San Isidro
- Poland (20):
  - Research Site, Bydgoszcz
  - Research Site, Gdansk
  - Research Site, Kamieniec Ząbkowicki
  - Research Site, Koluszki
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Mrgowo
  - Research Site, Nakso Nad Noteci
  - Research Site, Opole
  - Research Site, Oława
  - Research Site, Poznan
  - Research Site, Przemyśl
  - Research Site, Sieradz
  - Research Site, Skierniewice
  - Research Site, Torun
  - Research Site, Warsaw
  - Research Site, Wąbrzeźno
  - Research Site, Wroclaw
  - Research Site, Zabrze
  - Research Site, Łęczna
- Puerto Rico (10):
  - Research Site, Aguas Buneas
  - Research Site, Bayamón
  - Research Site, Cidra
  - Research Site, Hato Rey
  - Research Site, Jardines de Loiza, Loiza
  - Research Site, Juncos
  - Research Site, Ponce
  - Research Site, Rio Piedras
  - Research Site, San Juan
  - Research Site, Toa Baja
- Russia (7):
  - Research Site, Kazan'
  - Research Site, Moscow
  - Research Site, Novosibirsk
  - Research Site, Saint Petersburg
  - Research Site, Saratov
  - Research Site, StPetersburg
  - Research Site, Yekaterinburg
- South Africa (8):
  - Research Site, Benoni
  - Research Site, Cape Town
  - Research Site, Durban
  - Research Site, eMkhomazi
  - Research Site, Johannesburg
  - Research Site, Parow
  - Research Site, Pretoria
  - Research Site, Verulam
- Spain (12):
  - Research Site, Alicante
  - Research Site, Barcelona
  - Research Site, Granada
  - Research Site, Jerez de La Frontera Cadiz
  - Research Site, Lleida
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Oviedo
  - Research Site, Palma de Mallorca
  - Research Site, Santiago de Compostela
  - Research Site, Seville
  - Research Site, Valencia
- Sweden (12):
  - Research Site, Brämhult
  - Research Site, Eksjö
  - Research Site, Gothenburg
  - Research Site, Helsingborg
  - Research Site, Jönköping
  - Research Site, Malmo
  - Research Site, Örebro
  - Research Site, Östersund
  - Research Site, Rättvik
  - Research Site, Söråker
  - Research Site, Stockholm
  - Research Site, Umeå
- Taiwan (5):
  - Research Site, Kaohsiung City
  - Research Site, Kaohsiung Hsien
  - Research Site, Taichung
  - Research Site, Taipei
  - Research Site, Yongkang District
- Thailand (5):
  - Research Site, Bangkok
  - Research Site, Bangkoknoi
  - Research Site, Chiang Mai
  - Research Site, Khon Kaen
  - Research Site, Ratchaburi
- United Kingdom (17):
  - Research Site, Aylesbury
  - Research Site, Bath
  - Research Site, Belfast
  - Research Site, Blackpool
  - Research Site, Corsham
  - Research Site, Coventry
  - Research Site, Fowey
  - Research Site, Kenton
  - Research Site, Leicester
  - Research Site, Mortimer Reading
  - Research Site, Plymouth
  - Research Site, Sheffield
  - Research Site, Sunbury-on-Thames
  - Research Site, Swindon
  - Research Site, Wansford
  - Research Site, Warminster
  - Research Site, Whitstable

REFERENCES:
- [Derived] Cavallari I, Bhatt DL, Steg PG, Leiter LA, McGuire DK, Mosenzon O, Im K, Raz I, Braunwald E, Scirica BM. Causes and Risk Factors for Death in Diabetes: A Competing-Risk Analysis From the SAVOR-TIMI 53 Trial. J Am Coll Cardiol. 2021 Apr 13;77(14):1837-1840. doi: 10.1016/j.jacc.2021.02.030. No abstract available. PMID 33832610
- [Derived] Berg DD, Wiviott SD, Scirica BM, Gurmu Y, Mosenzon O, Murphy SA, Bhatt DL, Leiter LA, McGuire DK, Wilding JPH, Johanson P, Johansson PA, Langkilde AM, Raz I, Braunwald E, Sabatine MS. Heart Failure Risk Stratification and Efficacy of Sodium-Glucose Cotransporter-2 Inhibitors in Patients With Type 2 Diabetes Mellitus. Circulation. 2019 Nov 5;140(19):1569-1577. doi: 10.1161/CIRCULATIONAHA.119.042685. Epub 2019 Aug 31. PMID 31474116
- [Derived] Bergmark BA, Bhatt DL, McGuire DK, Cahn A, Mosenzon O, Steg PG, Im K, Kanevsky E, Gurmu Y, Raz I, Braunwald E, Scirica BM; SAVOR-TIMI 53 Steering Committee and Investigators. Metformin Use and Clinical Outcomes Among Patients With Diabetes Mellitus With or Without Heart Failure or Kidney Dysfunction: Observations From the SAVOR-TIMI 53 Trial. Circulation. 2019 Sep 17;140(12):1004-1014. doi: 10.1161/CIRCULATIONAHA.119.040144. Epub 2019 Jul 31. PMID 31362530
- [Derived] Scirica BM, Mosenzon O, Bhatt DL, Udell JA, Steg PG, McGuire DK, Im K, Kanevsky E, Stahre C, Sjostrand M, Raz I, Braunwald E. Cardiovascular Outcomes According to Urinary Albumin and Kidney Disease in Patients With Type 2 Diabetes at High Cardiovascular Risk: Observations From the SAVOR-TIMI 53 Trial. JAMA Cardiol. 2018 Feb 1;3(2):155-163. doi: 10.1001/jamacardio.2017.4228. PMID 29214305
- [Derived] Xia C, Goud A, D'Souza J, Dahagam C, Rao X, Rajagopalan S, Zhong J. DPP4 inhibitors and cardiovascular outcomes: safety on heart failure. Heart Fail Rev. 2017 May;22(3):299-304. doi: 10.1007/s10741-017-9617-4. PMID 28417296
- [Derived] Mosenzon O, Leibowitz G, Bhatt DL, Cahn A, Hirshberg B, Wei C, Im K, Rozenberg A, Yanuv I, Stahre C, Ray KK, Iqbal N, Braunwald E, Scirica BM, Raz I. Effect of Saxagliptin on Renal Outcomes in the SAVOR-TIMI 53 Trial. Diabetes Care. 2017 Jan;40(1):69-76. doi: 10.2337/dc16-0621. Epub 2016 Oct 17. PMID 27797925
- [Derived] Scirica BM, Bhatt DL, Braunwald E, Raz I, Cavender MA, Im K, Mosenzon O, Udell JA, Hirshberg B, Pollack PS, Steg PG, Jarolim P, Morrow DA. Prognostic Implications of Biomarker Assessments in Patients With Type 2 Diabetes at High Cardiovascular Risk: A Secondary Analysis of a Randomized Clinical Trial. JAMA Cardiol. 2016 Dec 1;1(9):989-998. doi: 10.1001/jamacardio.2016.3030. PMID 27681000
- [Derived] Cavender MA, Scirica BM, Raz I, Steg PG, McGuire DK, Leiter LA, Hirshberg B, Davidson J, Cahn A, Mosenzon O, Im K, Braunwald E, Bhatt DL. Cardiovascular Outcomes of Patients in SAVOR-TIMI 53 by Baseline Hemoglobin A1c. Am J Med. 2016 Mar;129(3):340.e1-8. doi: 10.1016/j.amjmed.2015.09.022. Epub 2015 Oct 31. PMID 26524706
- [Derived] Mosenzon O, Wei C, Davidson J, Scirica BM, Yanuv I, Rozenberg A, Hirshberg B, Cahn A, Stahre C, Strojek K, Bhatt DL, Raz I. Incidence of Fractures in Patients With Type 2 Diabetes in the SAVOR-TIMI 53 Trial. Diabetes Care. 2015 Nov;38(11):2142-50. doi: 10.2337/dc15-1068. Epub 2015 Sep 10. PMID 26358285
- [Derived] Leiter LA, Teoh H, Braunwald E, Mosenzon O, Cahn A, Kumar KM, Smahelova A, Hirshberg B, Stahre C, Frederich R, Bonnici F, Scirica BM, Bhatt DL, Raz I; SAVOR-TIMI 53 Steering Committee and Investigators. Efficacy and safety of saxagliptin in older participants in the SAVOR-TIMI 53 trial. Diabetes Care. 2015 Jun;38(6):1145-53. doi: 10.2337/dc14-2868. Epub 2015 Mar 10. PMID 25758769
- [Derived] Udell JA, Bhatt DL, Braunwald E, Cavender MA, Mosenzon O, Steg PG, Davidson JA, Nicolau JC, Corbalan R, Hirshberg B, Frederich R, Im K, Umez-Eronini AA, He P, McGuire DK, Leiter LA, Raz I, Scirica BM; SAVOR-TIMI 53 Steering Committee and Investigators. Saxagliptin and cardiovascular outcomes in patients with type 2 diabetes and moderate or severe renal impairment: observations from the SAVOR-TIMI 53 Trial. Diabetes Care. 2015 Apr;38(4):696-705. doi: 10.2337/dc14-1850. Epub 2014 Dec 31. PMID 25552421
- [Derived] Scirica BM, Braunwald E, Raz I, Cavender MA, Morrow DA, Jarolim P, Udell JA, Mosenzon O, Im K, Umez-Eronini AA, Pollack PS, Hirshberg B, Frederich R, Lewis BS, McGuire DK, Davidson J, Steg PG, Bhatt DL; SAVOR-TIMI 53 Steering Committee and Investigators*. Heart failure, saxagliptin, and diabetes mellitus: observations from the SAVOR-TIMI 53 randomized trial. Circulation. 2014 Oct 28;130(18):1579-88. doi: 10.1161/CIRCULATIONAHA.114.010389. Epub 2014 Sep 4. PMID 25189213
- [Derived] Scirica BM, Bhatt DL, Braunwald E, Steg PG, Davidson J, Hirshberg B, Ohman P, Frederich R, Wiviott SD, Hoffman EB, Cavender MA, Udell JA, Desai NR, Mosenzon O, McGuire DK, Ray KK, Leiter LA, Raz I; SAVOR-TIMI 53 Steering Committee and Investigators. Saxagliptin and cardiovascular outcomes in patients with type 2 diabetes mellitus. N Engl J Med. 2013 Oct 3;369(14):1317-26. doi: 10.1056/NEJMoa1307684. Epub 2013 Sep 2. PMID 23992601
- [Derived] Mosenzon O, Raz I, Scirica BM, Hirshberg B, Stahre CI, Steg PG, Davidson J, Ohman P, Price DL, Frederich B, Udell JA, Braunwald E, Bhatt DL. Baseline characteristics of the patient population in the Saxagliptin Assessment of Vascular Outcomes Recorded in patients with diabetes mellitus (SAVOR)-TIMI 53 trial. Diabetes Metab Res Rev. 2013 Jul;29(5):417-26. doi: 10.1002/dmrr.2413. Epub 2013 May 21. PMID 23564755
- [Derived] Scirica BM, Bhatt DL, Braunwald E, Steg PG, Davidson J, Hirshberg B, Ohman P, Price DL, Chen R, Udell J, Raz I. The design and rationale of the saxagliptin assessment of vascular outcomes recorded in patients with diabetes mellitus-thrombolysis in myocardial infarction (SAVOR-TIMI) 53 study. Am Heart J. 2011 Nov;162(5):818-825.e6. doi: 10.1016/j.ahj.2011.08.006. PMID 22093196
- See also: D1680C00003 Clinical Study Protocol — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=1185&filename=D1680C00003_CSP.pdf
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1185&filename=D1680C00003_Study_Synopsis_for_CTW.pdf
- See also: D1680C00003_CSR_Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1185&filename=D1680C00003_Study_Synopsis.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant was enrolled on 10 May 2010 and the last participant completed the study on 16 May 2013. A total of 18206 subjects were enrolled in the study of which 16492 were randomised. Study participants were randomized from 790 centers in 26 countries.
Pre-assignment Details: Subjects meeting all inclusion criteria and with no exclusion criteria were randomised in a 1:1 ratio to receive either saxagliptin or matching placebo (Day 0).
Groups:
- Saxagliptin: 5 mg once daily in subjects with normal renal function or mild impaired renal function (eGFR >50 mL/min); 2.5 mg once daily in subjects with moderate to severe renal impairment (eGFR ≤50 mL/min).
- Placebo: Matching Placebo
Period: Overall Study
Arm/Group | Saxagliptin | Placebo
Started | 8280 (Randomized subjects) | 8212 (Randomized subjects)
Completed | 8078 (Completed subjects) | 7998 (Completed subjects)
Not Completed | 202 | 214
Not completed — Lost to Follow-up | 15 | 13
Not completed — Withdrawal by Subject | 180 | 196
Not completed — Administrative withdrawal of consent | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saxagliptin | Placebo | Total
Number analyzed (Participants) | 8280 | 8212 | 16492
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.1 (8.52) | 65.0 (8.58) | 65.0 (8.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2768 | 2687 | 5455
  Male | 5512 | 5525 | 11037
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1778 | 1763 | 3541
  Not Hispanic or Latino | 6502 | 6449 | 12951
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 18 | 33 | 51
  Asian | 896 | 884 | 1780
  Native Hawaiian or Other Pacific Islander | 11 | 11 | 22
  Black or African American | 278 | 290 | 568
  White | 6241 | 6166 | 12407
  More than one race | 768 | 758 | 1526
  Unknown or Not Reported | 68 | 70 | 138
Cardiovascular Risk Category: Cardiovascular disease/Multiple risk factors (CVD/MRF) [Number; unit: Participants] — CVD subjects were defined as subjects with history of established CV disease. MRF subjects were defined as subjects with MRF for vascular disease without established CV disease.
  Participants
    CVD | 6494 | 6465 | 12959
    MRF | 1786 | 1747 | 3533
Renal Functione Categor: Normal or Mild impairment/Moderate impairment/Severe impairment [Number; unit: Participants] — Renal function categories Normal function - Mild impairment defined as: eGFR >50 mL/min; Moderate impairment defined as: eGFR 30 to 50 mL/min; Severe impairment defined as: eGFR eGFR <30 mL/min.
  Participants
    Normal or Mild impairment | 6986 | 6930 | 13916
    Moderate impairment | 1122 | 1118 | 2240
    Severe impairment | 172 | 164 | 336

OUTCOME MEASURES:

1. Primary Outcome: Participants With Any Event From the Composite of Cardiovascular Death (CV Death), Non-fatal Myocardial Infarction (MI), or Non-fatal Ischaemic Stroke
Description: Participants with CV death, non-fatal MI or non-fatal ischaemic stroke. If no event, censoring occurs at the patient withdrawal of consent, last contact, or death (when applicable)-whichever was later.
Time Frame: Randomization (day 0) up to 2.9 years
Population: Intention To Treat (ITT) analysis of randomized population. Events were adjudicated by the Clinical Event Adjudication Committee.
Measure: Number; unit: participants
Arm/Group | Saxagliptin | Placebo
Number analyzed (Participants) | 8280 | 8212
participants | 613 | 609

2. Secondary Outcome: Participants With Any Event From the Composite of CV Death, Non-fatal MI, Non-fatal Ischaemic Stroke, Hospitalisation for Heart Failure, Hospitalisation for Unstable Angina Pectoris, or Hospitalisation for Coronary Revascularisation
Description: Participants with CV death, non-fatal MI, non-fatal ischaemic stroke, hospitalisation for heart failure, hospitalisation for unstable angina pectoris, or hospitalisation for coronary revascularisation. If no event, censoring occurs at the patient withdrawal of consent, last contact, or death (when applicable)-whichever was later.
Time Frame: Randomization (day 0) up to 2.9 years
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Saxagliptin | Placebo
Number analyzed (Participants) | 8280 | 8212
participants | 1059 | 1034

3. Secondary Outcome: Participants With Event of Death
Description: Participants with event of death. If no event, censoring occurs at the patient withdrawal of consent, or last contact -whichever was later.
Time Frame: Randomization (day 0) up to 2.9 years
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Saxagliptin | Placebo
Number analyzed (Participants) | 8280 | 8212
participants | 420 | 378

ADVERSE EVENTS:
Arm/Group | Placebo | Saxagliptin
Serious Adverse Events (participants affected / at risk) | 2075/8212 | 2114/8280
Other Adverse Events (participants affected / at risk) | 3641/8212 | 3504/8280
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=8212) | Saxagliptin (N=8280)
Anaemia (Blood and lymphatic system disorders) | 26 (27) | 17 (19)
Anaemia megaloblastic (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypereosinophilic syndrome (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypochromic anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 7 (7) | 5 (5)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 4 (4)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Pernicious anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 5 (5)
Acute coronary syndrome (Cardiac disorders) | 7 (7) | 5 (5)
Acute left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 6 (6)
Adams-Stokes syndrome (Cardiac disorders) | 0 (0) | 2 (2)
Angina pectoris (Cardiac disorders) | 106 (116) | 89 (98)
Angina unstable (Cardiac disorders) | 63 (79) | 44 (48)
Aortic valve stenosis (Cardiac disorders) | 5 (5) | 6 (6)
Arrhythmia (Cardiac disorders) | 4 (4) | 3 (3)
Arteriosclerosis coronary artery (Cardiac disorders) | 2 (2) | 2 (2)
Arteriospasm coronary (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 76 (90) | 78 (85)
Atrial flutter (Cardiac disorders) | 11 (13) | 22 (25)
Atrial septal defect acquired (Cardiac disorders) | 1 (1) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Atrial thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block (Cardiac disorders) | 3 (3) | 3 (3)
Atrioventricular block complete (Cardiac disorders) | 13 (13) | 6 (6)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 5 (6) | 2 (2)
Bifascicular block (Cardiac disorders) | 0 (0) | 1 (1)
Bradyarrhythmia (Cardiac disorders) | 4 (4) | 0 (0)
Bradycardia (Cardiac disorders) | 11 (11) | 14 (15)
Bundle branch block (Cardiac disorders) | 0 (0) | 1 (1)
Bundle branch block left (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac aneurysm (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 4 (4) | 5 (5)
Cardiac failure (Cardiac disorders) | 24 (24) | 21 (22)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 3 (3)
Cardiac failure chronic (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 21 (22) | 30 (30)
Cardiac fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 2 (2)
Cardiac valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 3 (3) | 2 (2)
Cardiopulmonary failure (Cardiac disorders) | 2 (2) | 0 (0)
Cardiovascular disorder (Cardiac disorders) | 0 (0) | 1 (1)
Cardiovascular insufficiency (Cardiac disorders) | 0 (0) | 1 (1)
Congestive cardiomyopathy (Cardiac disorders) | 2 (2) | 2 (2)
Cor pulmonale (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 18 (19) | 17 (17)
Coronary artery insufficiency (Cardiac disorders) | 2 (2) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 2 (2) | 0 (0)
Diastolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Hypertensive heart disease (Cardiac disorders) | 1 (1) | 1 (1)
Hypertrophic cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Intracardiac thrombus (Cardiac disorders) | 2 (2) | 2 (2)
Ischaemic cardiomyopathy (Cardiac disorders) | 6 (7) | 3 (3)
Left ventricular dysfunction (Cardiac disorders) | 3 (3) | 1 (1)
Left ventricular failure (Cardiac disorders) | 0 (0) | 2 (3)
Mitral valve incompetence (Cardiac disorders) | 3 (3) | 3 (3)
Myocardial infarction (Cardiac disorders) | 5 (5) | 3 (3)
Myocardial ischaemia (Cardiac disorders) | 11 (11) | 7 (7)
Nodal arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 4 (4) | 3 (3)
Pericardial effusion (Cardiac disorders) | 1 (1) | 2 (2)
Pericarditis (Cardiac disorders) | 3 (4) | 0 (0)
Pulseless electrical activity (Cardiac disorders) | 1 (1) | 0 (0)
Right ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 14 (14) | 10 (10)
Sinoatrial block (Cardiac disorders) | 1 (1) | 0 (0)
Sinus arrhythmia (Cardiac disorders) | 2 (2) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 6 (6) | 3 (3)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 4 (4) | 9 (10)
Systolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Tachyarrhythmia (Cardiac disorders) | 1 (2) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (3) | 8 (8)
Torsade de pointes (Cardiac disorders) | 1 (1) | 0 (0)
Tricuspid valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Trifascicular block (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 2 (2) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 4 (4) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 5 (5) | 3 (3)
Ventricular hypokinesia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 11 (16) | 16 (17)
Deafness (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Meniere's disease (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Sudden hearing loss (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (2)
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 (0) | 1 (2)
Vertigo (Ear and labyrinth disorders) | 10 (10) | 16 (16)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 3 (3)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 1 (1) | 2 (2)
Hypercorticoidism (Endocrine disorders) | 1 (1) | 0 (0)
Hyperparathyroidism primary (Endocrine disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 2 (2) | 6 (6)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Toxic nodular goitre (Endocrine disorders) | 0 (0) | 1 (1)
Angle closure glaucoma (Eye disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 13 (15) | 7 (9)
Cataract cortical (Eye disorders) | 0 (0) | 1 (1)
Diabetic retinopathy (Eye disorders) | 1 (1) | 6 (7)
Diplopia (Eye disorders) | 1 (1) | 1 (1)
Eye haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 2 (2)
Macular oedema (Eye disorders) | 0 (0) | 1 (1)
Optic ischaemic neuropathy (Eye disorders) | 3 (3) | 0 (0)
Retinal artery occlusion (Eye disorders) | 1 (1) | 1 (1)
Retinal detachment (Eye disorders) | 2 (2) | 1 (1)
Retinal haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Retinal ischaemia (Eye disorders) | 0 (0) | 1 (1)
Ulcerative keratitis (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 2 (2)
Vitreous haemorrhage (Eye disorders) | 3 (3) | 2 (2)
Abdominal adhesions (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 5 (5) | 3 (3)
Abdominal hernia obstructive (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 13 (14) | 17 (17)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 4 (4)
Abdominal strangulated hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal wall haematoma (Gastrointestinal disorders) | 3 (3) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 2 (3) | 0 (0)
Anal polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 4 (4) | 3 (3)
Colitis (Gastrointestinal disorders) | 5 (5) | 4 (4)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 6 (6)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colonic polyp (Gastrointestinal disorders) | 4 (4) | 6 (6)
Colonic pseudo-obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (5) | 4 (4)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diabetic gastroparesis (Gastrointestinal disorders) | 2 (5) | 1 (1)
Diaphragmatic hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 15 (15) | 12 (13)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulitis intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum oesophageal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 7 (7) | 4 (4)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 2 (2) | 2 (2)
Duodenal ulcer perforation (Gastrointestinal disorders) | 3 (3) | 0 (0)
Dyskinesia oesophageal (Gastrointestinal disorders) | 1 (3) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 3 (3)
Enteritis (Gastrointestinal disorders) | 0 (0) | 3 (3)
Enterovesical fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Femoral hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastric antral vascular ectasia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 4 (4) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 7 (7) | 3 (3)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 4 (4) | 3 (3)
Gastritis (Gastrointestinal disorders) | 11 (12) | 15 (15)
Gastritis atrophic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 3 (3) | 1 (1)
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 18 (25) | 15 (15)
Gastrointestinal hypomotility (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrointestinal telangiectasia (Gastrointestinal disorders) | 3 (3) | 0 (0)
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal vascular malformation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 8 (8) | 7 (7)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Haematochezia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 4 (4) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 3 (3) | 5 (5)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Ileus (Gastrointestinal disorders) | 1 (1) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inflammatory bowel disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 4 (4) | 6 (6)
Inguinal hernia, obstructive (Gastrointestinal disorders) | 2 (2) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 2 (3) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 3 (3) | 5 (5)
Intestinal perforation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Intestinal polyp haemorrhage (Gastrointestinal disorders) | 3 (3) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 1 (1)
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 (4) | 0 (0)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 (0) | 2 (2)
Megacolon (Gastrointestinal disorders) | 1 (1) | 1 (1)
Mesenteric artery stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mesenteric artery thrombosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mesenteric vascular insufficiency (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 4 (4)
Oesophageal fibrosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal spasm (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 4 (4)
Oesophagitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1)
Omental infarction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic duct dilatation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic mass (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 12 (14) | 18 (19)
Pancreatitis acute (Gastrointestinal disorders) | 6 (6) | 4 (5)
Pancreatitis chronic (Gastrointestinal disorders) | 2 (2) | 2 (2)
Pancreatolithiasis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Rectal polyp (Gastrointestinal disorders) | 2 (2) | 2 (2)
Rectal prolapse (Gastrointestinal disorders) | 0 (0) | 3 (3)
Reflux gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Retroperitoneal fibrosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 4 (6) | 4 (4)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 3 (3)
Tongue disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 4 (4) | 5 (5)
Umbilical hernia, obstructive (Gastrointestinal disorders) | 2 (2) | 3 (3)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 9 (10) | 5 (5)
Varices oesophageal (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 6 (6)
Adverse drug reaction (General disorders) | 2 (2) | 1 (1)
Application site pain (General disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 4 (4)
Catheter site haemorrhage (General disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 2 (3) | 0 (0)
Chest pain (General disorders) | 10 (10) | 14 (14)
Cyst (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 5 (5)
Device battery issue (General disorders) | 1 (1) | 0 (0)
Device breakage (General disorders) | 0 (0) | 3 (3)
Device damage (General disorders) | 0 (0) | 1 (1)
Device dislocation (General disorders) | 1 (1) | 1 (1)
Device failure (General disorders) | 1 (1) | 1 (1)
Device lead damage (General disorders) | 1 (1) | 1 (1)
Device malfunction (General disorders) | 0 (0) | 4 (4)
Exercise tolerance decreased (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 3 (3)
Feeling cold (General disorders) | 0 (0) | 1 (1)
Foaming at mouth (General disorders) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 2 (2) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 1 (1)
General symptom (General disorders) | 0 (0) | 1 (1)
Generalised oedema (General disorders) | 2 (2) | 1 (1)
Hernia (General disorders) | 0 (0) | 1 (1)
Hernia obstructive (General disorders) | 0 (0) | 1 (1)
Hypothermia (General disorders) | 1 (1) | 0 (0)
Impaired healing (General disorders) | 1 (1) | 3 (3)
Implant site haematoma (General disorders) | 1 (1) | 0 (0)
Inflammation (General disorders) | 1 (1) | 2 (2)
Ischaemic ulcer (General disorders) | 1 (2) | 0 (0)
Lipogranuloma (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0)
Medical device complication (General disorders) | 0 (0) | 1 (1)
Multi-organ disorder (General disorders) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 5 (5) | 7 (7)
Necrobiosis (General disorders) | 0 (0) | 1 (1)
Necrosis (General disorders) | 0 (0) | 1 (2)
Non-cardiac chest pain (General disorders) | 109 (131) | 108 (125)
Oedema peripheral (General disorders) | 1 (1) | 4 (4)
Organ failure (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 2 (2)
Polyp (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 7 (7) | 7 (7)
Spinal pain (General disorders) | 0 (0) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 3 (3)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 5 (5) | 3 (3)
Biliary colic (Hepatobiliary disorders) | 4 (4) | 0 (0)
Biliary dyskinesia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Biliary polyp (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholangitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 10 (12) | 13 (13)
Cholecystitis acute (Hepatobiliary disorders) | 14 (14) | 22 (22)
Cholecystitis chronic (Hepatobiliary disorders) | 4 (4) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 27 (28) | 26 (27)
Drug-induced liver injury (Hepatobiliary disorders) | 2 (2) | 0 (0)
Gallbladder disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gallbladder perforation (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 6 (6) | 2 (2)
Hepatic failure (Hepatobiliary disorders) | 2 (2) | 3 (3)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatic ischaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic lesion (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hydrocholecystis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Ischaemic hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 2 (2) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 2 (2) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Allergy to venom (Immune system disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 1 (1)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1)
Autoimmune disorder (Immune system disorders) | 0 (0) | 1 (1)
Cryoglobulinaemia (Immune system disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 4 (4) | 4 (4)
Hypersensitivity (Immune system disorders) | 0 (0) | 3 (3)
Sarcoidosis (Immune system disorders) | 1 (1) | 1 (1)
Abdominal abscess (Infections and infestations) | 1 (1) | 1 (1)
Abdominal wall abscess (Infections and infestations) | 1 (1) | 1 (1)
Abscess (Infections and infestations) | 2 (2) | 0 (0)
Abscess limb (Infections and infestations) | 4 (4) | 5 (5)
Abscess soft tissue (Infections and infestations) | 1 (1) | 0 (0)
Acarodermatitis (Infections and infestations) | 0 (0) | 1 (1)
Acinetobacter bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Adenovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 1 (2) | 0 (0)
Appendicitis (Infections and infestations) | 9 (9) | 7 (7)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 2 (2) | 3 (3)
Arthritis infective (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 2 (2) | 3 (3)
Bacterial infection (Infections and infestations) | 1 (1) | 1 (1)
Bacterial sepsis (Infections and infestations) | 1 (1) | 1 (1)
Bone abscess (Infections and infestations) | 0 (0) | 1 (1)
Breast cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Breast infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 35 (35) | 23 (23)
Bronchitis viral (Infections and infestations) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 8 (9) | 10 (10)
Bursitis infective (Infections and infestations) | 1 (1) | 0 (0)
Campylobacter infection (Infections and infestations) | 0 (0) | 1 (1)
Carbuncle (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 65 (70) | 58 (70)
Cellulitis gangrenous (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis of male external genital organ (Infections and infestations) | 1 (1) | 1 (1)
Cellulitis staphylococcal (Infections and infestations) | 3 (3) | 1 (1)
Cervicitis (Infections and infestations) | 0 (0) | 1 (1)
Chest wall abscess (Infections and infestations) | 1 (1) | 0 (0)
Cholangitis suppurative (Infections and infestations) | 0 (0) | 1 (1)
Cholecystitis infective (Infections and infestations) | 1 (1) | 0 (0)
Chronic sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Clostridial infection (Infections and infestations) | 0 (0) | 2 (2)
Clostridium difficile colitis (Infections and infestations) | 6 (6) | 2 (2)
Clostridium difficile sepsis (Infections and infestations) | 1 (1) | 0 (0)
Creutzfeldt-Jakob disease (Infections and infestations) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 2 (2) | 2 (4)
Dengue fever (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 2 (2) | 2 (2)
Diabetic foot infection (Infections and infestations) | 3 (3) | 10 (11)
Diabetic gangrene (Infections and infestations) | 4 (4) | 9 (9)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 10 (13) | 10 (11)
Ear infection (Infections and infestations) | 0 (0) | 1 (1)
Emphysematous cystitis (Infections and infestations) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1) | 1 (1)
Endocarditis enterococcal (Infections and infestations) | 0 (0) | 1 (1)
Endophthalmitis (Infections and infestations) | 1 (1) | 0 (0)
Enterobacter bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Enterobacter infection (Infections and infestations) | 1 (1) | 0 (0)
Enterobacter pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Enterococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 2 (2)
Erysipelas (Infections and infestations) | 6 (6) | 6 (6)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 1 (1)
Escherichia infection (Infections and infestations) | 1 (1) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Febrile infection (Infections and infestations) | 1 (1) | 0 (0)
Furuncle (Infections and infestations) | 1 (1) | 0 (0)
Gallbladder abscess (Infections and infestations) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 16 (17) | 22 (23)
Gastric ulcer helicobacter (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 17 (17) | 28 (29)
Gastroenteritis clostridial (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis norovirus (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis shigella (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 3 (3)
Graft infection (Infections and infestations) | 3 (3) | 0 (0)
Groin abscess (Infections and infestations) | 1 (1) | 0 (0)
Groin infection (Infections and infestations) | 1 (1) | 0 (0)
H1N1 influenza (Infections and infestations) | 1 (1) | 1 (1)
HIV infection (Infections and infestations) | 0 (0) | 1 (1)
Helicobacter infection (Infections and infestations) | 3 (3) | 1 (1)
Hepatitis B (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1)
Herpes zoster ophthalmic (Infections and infestations) | 1 (1) | 0 (0)
Implant site cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Incision site infection (Infections and infestations) | 1 (1) | 0 (0)
Infected dermal cyst (Infections and infestations) | 1 (1) | 0 (0)
Infected fistula (Infections and infestations) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 8 (9) | 4 (4)
Infection (Infections and infestations) | 1 (1) | 3 (3)
Infectious peritonitis (Infections and infestations) | 2 (2) | 0 (0)
Infectious thyroiditis (Infections and infestations) | 1 (1) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 2 (2) | 6 (6)
Intestinal gangrene (Infections and infestations) | 0 (0) | 1 (1)
Klebsiella infection (Infections and infestations) | 0 (0) | 1 (1)
Labyrinthitis (Infections and infestations) | 1 (1) | 1 (1)
Liver abscess (Infections and infestations) | 2 (2) | 1 (1)
Lobar pneumonia (Infections and infestations) | 8 (8) | 16 (16)
Localised infection (Infections and infestations) | 11 (11) | 8 (8)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 4 (6)
Ludwig angina (Infections and infestations) | 1 (1) | 0 (0)
Lung infection pseudomonal (Infections and infestations) | 1 (1) | 0 (0)
Lyme disease (Infections and infestations) | 0 (0) | 1 (1)
Mastoiditis (Infections and infestations) | 1 (1) | 0 (0)
Mediastinitis (Infections and infestations) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 1 (1)
Necrotising fasciitis (Infections and infestations) | 4 (4) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Orchitis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 24 (25) | 18 (23)
Osteomyelitis chronic (Infections and infestations) | 3 (3) | 0 (0)
Otitis externa (Infections and infestations) | 1 (1) | 2 (2)
Parametritis (Infections and infestations) | 0 (0) | 1 (1)
Pelvic abscess (Infections and infestations) | 1 (1) | 0 (0)
Peridiverticular abscess (Infections and infestations) | 1 (1) | 0 (0)
Perihepatic abscess (Infections and infestations) | 0 (0) | 1 (1)
Perineal abscess (Infections and infestations) | 1 (1) | 1 (1)
Perinephric abscess (Infections and infestations) | 0 (0) | 1 (1)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Perirectal abscess (Infections and infestations) | 1 (1) | 0 (0)
Peritoneal abscess (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 4 (4) | 5 (5)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pilonidal cyst (Infections and infestations) | 2 (2) | 0 (0)
Pneumococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Pneumococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Pneumocystis jiroveci infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 118 (127) | 151 (168)
Pneumonia bacterial (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia chlamydial (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia fungal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia legionella (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia mycoplasmal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 2 (2) | 3 (3)
Post procedural sepsis (Infections and infestations) | 0 (0) | 1 (1)
Postoperative abscess (Infections and infestations) | 2 (2) | 2 (2)
Postoperative wound infection (Infections and infestations) | 9 (10) | 8 (9)
Prostatic abscess (Infections and infestations) | 0 (0) | 1 (1)
Pseudomonal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 4 (4) | 6 (6)
Pyelonephritis (Infections and infestations) | 7 (7) | 11 (11)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 5 (6)
Rectal abscess (Infections and infestations) | 1 (1) | 0 (0)
Renal abscess (Infections and infestations) | 0 (0) | 3 (3)
Respiratory tract infection (Infections and infestations) | 3 (3) | 2 (2)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 1 (1)
Retroperitoneal abscess (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 20 (22) | 21 (21)
Sepsis syndrome (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 9 (9) | 11 (11)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Skin bacterial infection (Infections and infestations) | 2 (2) | 0 (0)
Skin infection (Infections and infestations) | 1 (2) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 4 (4) | 3 (5)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal skin infection (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 1 (1) | 1 (1)
Streptococcal urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 3 (3) | 4 (4)
Subdiaphragmatic abscess (Infections and infestations) | 0 (0) | 1 (1)
Syphilis (Infections and infestations) | 1 (1) | 0 (0)
Testicular abscess (Infections and infestations) | 0 (0) | 1 (1)
Thrombophlebitis septic (Infections and infestations) | 0 (0) | 1 (1)
Tracheobronchitis (Infections and infestations) | 1 (1) | 1 (1)
Typhoid fever (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 7 (7) | 7 (8)
Urinary tract infection (Infections and infestations) | 49 (50) | 40 (42)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 8 (8) | 10 (10)
Vaginal abscess (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 4 (4) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Vulval abscess (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 7 (7) | 7 (7)
Wound infection staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Wound sepsis (Infections and infestations) | 2 (2) | 1 (1)
Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Anastomotic ulcer haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 8 (8) | 3 (3)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Arteriovenous graft site haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bone fissure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Brachial plexus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Burns second degree (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Burns third degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cartilage injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 2 (2) | 5 (5)
Contrast media reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Craniocerebral injury (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Cystitis radiation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 8 (8) | 6 (6)
Feeding tube complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 5 (5) | 10 (10)
Femur fracture (Injury, poisoning and procedural complications) | 10 (10) | 13 (15)
Fibula fracture (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Foreign body (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fractured coccyx (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Graft complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Graft dysfunction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Graft thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 1 (2)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Head injury (Injury, poisoning and procedural complications) | 4 (4) | 5 (5)
Heart injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 10 (10) | 8 (9)
Humerus fracture (Injury, poisoning and procedural complications) | 5 (5) | 9 (9)
Incisional hernia (Injury, poisoning and procedural complications) | 5 (5) | 6 (6)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Laceration (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 2 (2) | 7 (7)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Meniscus lesion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Multiple drug overdose intentional (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Near drowning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 5 (5)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Peripheral artery restenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post concussion syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post embolisation syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural bile leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Post procedural discharge (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 5 (6) | 1 (1)
Postoperative fever (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Postoperative hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative renal failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1) | 5 (5)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Pubis fracture (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Radius fracture (Injury, poisoning and procedural complications) | 5 (5) | 5 (5)
Rib fracture (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)
Road traffic accident (Injury, poisoning and procedural complications) | 7 (7) | 4 (4)
Scapula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Skeletal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skull fractured base (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 7 (7) | 2 (2)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Splenic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Splenic rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sternal fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 8 (8) | 9 (9)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Suture related complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 5 (5) | 5 (5)
Tracheal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic ulcer (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Vascular graft complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound necrosis (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Wound secretion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 3 (3) | 6 (6)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Arteriogram coronary (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 2 (2) | 1 (1)
Blood glucose increased (Investigations) | 1 (1) | 0 (0)
Blood potassium increased (Investigations) | 1 (1) | 0 (0)
Blood pressure abnormal (Investigations) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 2 (2) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1)
Cardiac stress test abnormal (Investigations) | 1 (1) | 1 (1)
Chest X-ray abnormal (Investigations) | 1 (1) | 0 (0)
Clostridium test positive (Investigations) | 1 (1) | 1 (1)
Coagulation factor VIII level increased (Investigations) | 1 (1) | 0 (0)
Coagulation test abnormal (Investigations) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 3 (3) | 0 (0)
Electrocardiogram abnormal (Investigations) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Heart rate increased (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 6 (6) | 5 (5)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1)
Liver function test abnormal (Investigations) | 3 (3) | 2 (2)
Prostatic specific antigen increased (Investigations) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 4 (4)
Troponin increased (Investigations) | 1 (1) | 1 (1)
Urine albumin/creatinine ratio increased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 17 (18) | 13 (13)
Diabetes mellitus (Metabolism and nutrition disorders) | 13 (14) | 12 (14)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 11 (13) | 10 (12)
Diabetic complication (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 5 (6) | 8 (10)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 5 (5) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 2 (2) | 8 (8)
Hypercalcaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 58 (62) | 51 (55)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 13 (15) | 17 (17)
Hyperosmolar state (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 7 (8) | 3 (3)
Hypovolaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Lactic acidosis (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 8 (8)
Arthritis (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Articular calcification (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (10) | 9 (9)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5)
Carpal collapse (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Diabetic amyotrophy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Extraskeletal ossification (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hip deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Inguinal mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (5)
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 13 (14) | 9 (10)
Joint ankylosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 3 (3) | 6 (6)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Monarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 32 (35) | 23 (23)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 40 (42) | 49 (51)
Osteochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 8 (8)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Polymyositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Spinal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 6 (6) | 7 (7)
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Vertebral column mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (4) | 0 (0)
Adenocarcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Angiocentric lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 42 (57) | 52 (58)
Basosquamous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Benign neoplasm of choroid (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (9) | 12 (13)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 2 (2)
Bladder cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Bladder transitional cell carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Blast crisis in myelogenous leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bone neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 (12) | 10 (10)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4)
Burkitt's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Carcinoid tumour of the gastrointestinal tract (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Central nervous system lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Choroid melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (3)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 18 (18) | 13 (13)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (4)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2)
Endometrial cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gallbladder cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (11) | 6 (6)
Gastric cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Head and neck cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 7 (7)
Hepatic neoplasm malignant recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hodgkin's disease nodular sclerosis stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Laryngeal cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Lip neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 2 (2)
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Lung adenocarcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 6 (6)
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung carcinoma cell type unspecified stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung carcinoma cell type unspecified stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 6 (6)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 15 (16) | 19 (20)
Lung squamous cell carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 5 (5)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (9) | 11 (11)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant palate neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant urinary tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Monoclonal gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Myeloproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Ocular neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Ovarian fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 2 (2)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic neuroendocrine tumour metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 34 (34) | 41 (43)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Prostate cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 0 (0)
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 4 (4)
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 4 (4)
Renal cell carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Retroperitoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rhabdomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Sarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Sinonasal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 5 (5)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 2 (2)
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1)
Small intestine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 30 (32) | 18 (19)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 7 (7)
Superficial spreading melanoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (7) | 1 (1)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Vascular neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Arachnoid cyst (Nervous system disorders) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1) | 1 (1)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1)
Basal ganglia haemorrhage (Nervous system disorders) | 1 (1) | 1 (1)
Brain injury (Nervous system disorders) | 0 (0) | 1 (1)
Brain mass (Nervous system disorders) | 1 (1) | 0 (0)
Brain stem haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Carotid arteriosclerosis (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery disease (Nervous system disorders) | 0 (0) | 3 (4)
Carotid artery occlusion (Nervous system disorders) | 1 (2) | 3 (3)
Carotid artery stenosis (Nervous system disorders) | 11 (11) | 29 (29)
Carotid sinus syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 3 (3) | 1 (2)
Cerebral arteriosclerosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral circulatory failure (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 2 (2) | 2 (2)
Cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral microangiopathy (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 14 (14) | 12 (12)
Cerebrovascular disorder (Nervous system disorders) | 2 (2) | 3 (3)
Cerebrovascular insufficiency (Nervous system disorders) | 1 (1) | 1 (1)
Cervical myelopathy (Nervous system disorders) | 1 (1) | 0 (0)
Cervical root pain (Nervous system disorders) | 0 (0) | 1 (1)
Cervicobrachial syndrome (Nervous system disorders) | 2 (2) | 1 (1)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0)
Coma (Nervous system disorders) | 1 (1) | 0 (0)
Complex partial seizures (Nervous system disorders) | 0 (0) | 2 (2)
Convulsion (Nervous system disorders) | 4 (4) | 3 (3)
Dementia (Nervous system disorders) | 0 (0) | 2 (3)
Dementia Alzheimer's type (Nervous system disorders) | 1 (1) | 0 (0)
Demyelinating polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Diabetic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 6 (6) | 7 (7)
Dizziness (Nervous system disorders) | 10 (11) | 16 (16)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Encephalitis (Nervous system disorders) | 1 (1) | 0 (0)
Encephalomalacia (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Epilepsy (Nervous system disorders) | 7 (8) | 2 (2)
Fahr's disease (Nervous system disorders) | 1 (1) | 0 (0)
Guillain-Barre syndrome (Nervous system disorders) | 1 (2) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 2 (2) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 4 (4)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Hemiparesis (Nervous system disorders) | 2 (2) | 4 (4)
Hemiplegia (Nervous system disorders) | 0 (0) | 1 (1)
Hemisensory neglect (Nervous system disorders) | 0 (0) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 2 (2) | 1 (1)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Hypertensive encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
IIIrd nerve paresis (Nervous system disorders) | 0 (0) | 1 (1)
IVth nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 1 (1)
Intraventricular haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 4 (4)
Lacunar infarction (Nervous system disorders) | 2 (2) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 2 (2) | 1 (1)
Mental impairment (Nervous system disorders) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Monoplegia (Nervous system disorders) | 0 (0) | 1 (1)
Movement disorder (Nervous system disorders) | 1 (1) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 1 (1) | 0 (0)
Nerve root compression (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (2) | 0 (0)
Neurological symptom (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 2 (2) | 2 (2)
Occipital neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Optic neuritis (Nervous system disorders) | 0 (0) | 1 (1)
Orthostatic intolerance (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 2 (2) | 2 (2)
Parkinson's disease (Nervous system disorders) | 1 (1) | 3 (3)
Parkinsonism (Nervous system disorders) | 0 (0) | 1 (1)
Polyneuropathy (Nervous system disorders) | 3 (3) | 0 (0)
Presyncope (Nervous system disorders) | 4 (4) | 5 (5)
Radicular pain (Nervous system disorders) | 1 (1) | 0 (0)
Radicular syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 2 (2) | 1 (1)
Sensory disturbance (Nervous system disorders) | 1 (1) | 0 (0)
Speech disorder (Nervous system disorders) | 1 (1) | 0 (0)
Spinal cord infarction (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 2 (2) | 4 (4)
Syncope (Nervous system disorders) | 32 (33) | 37 (39)
Tension headache (Nervous system disorders) | 0 (0) | 1 (1)
Thalamus haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 60 (64) | 48 (49)
Ulnar nerve palsy (Nervous system disorders) | 0 (0) | 1 (1)
Uraemic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
VIIth nerve paralysis (Nervous system disorders) | 4 (4) | 8 (8)
Vascular dementia (Nervous system disorders) | 1 (1) | 1 (1)
Vascular encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Vertebral artery stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Vertebrobasilar insufficiency (Nervous system disorders) | 3 (3) | 3 (3)
Vocal cord paralysis (Nervous system disorders) | 1 (1) | 0 (0)
White matter lesion (Nervous system disorders) | 0 (0) | 1 (1)
Adjustment disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Adjustment disorder with depressed mood (Psychiatric disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Alcoholism (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 3 (3)
Bipolar disorder (Psychiatric disorders) | 1 (2) | 2 (2)
Completed suicide (Psychiatric disorders) | 2 (2) | 1 (1)
Confusional state (Psychiatric disorders) | 2 (2) | 7 (8)
Delirium (Psychiatric disorders) | 1 (1) | 2 (2)
Depression (Psychiatric disorders) | 6 (8) | 5 (5)
Drug abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 1 (2) | 0 (0)
Mental status changes (Psychiatric disorders) | 5 (5) | 7 (8)
Psychosomatic disease (Psychiatric disorders) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 2 (2)
Stress (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 2 (2) | 0 (0)
Suicide attempt (Psychiatric disorders) | 4 (4) | 3 (3)
Acute prerenal failure (Renal and urinary disorders) | 1 (1) | 2 (2)
Azotaemia (Renal and urinary disorders) | 2 (2) | 3 (3)
Bladder outlet obstruction (Renal and urinary disorders) | 2 (2) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 2 (2) | 0 (0)
Calculus ureteric (Renal and urinary disorders) | 7 (8) | 5 (7)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 2 (2)
Cystitis haemorrhagic (Renal and urinary disorders) | 2 (2) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 1 (1)
Diabetic nephropathy (Renal and urinary disorders) | 0 (0) | 3 (3)
Glomerulonephritis membranoproliferative (Renal and urinary disorders) | 1 (1) | 0 (0)
Glomerulonephritis membranous (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 7 (7) | 5 (6)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 1 (1)
Lupus nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 11 (11) | 13 (16)
Nephropathy (Renal and urinary disorders) | 0 (0) | 2 (2)
Nephropathy toxic (Renal and urinary disorders) | 1 (1) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 3 (3) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 20 (20) | 23 (23)
Renal failure acute (Renal and urinary disorders) | 65 (71) | 80 (89)
Renal failure chronic (Renal and urinary disorders) | 17 (18) | 18 (19)
Renal impairment (Renal and urinary disorders) | 24 (25) | 22 (25)
Renal infarct (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal mass (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal tubular necrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Stress urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureteric stenosis (Renal and urinary disorders) | 2 (2) | 2 (2)
Urethral stenosis (Renal and urinary disorders) | 2 (2) | 5 (6)
Urinary bladder polyp (Renal and urinary disorders) | 0 (0) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 4 (4) | 8 (8)
Urinary tract obstruction (Renal and urinary disorders) | 4 (4) | 0 (0)
Acquired hydrocele (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Acquired phimosis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Balanitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 13 (13) | 13 (13)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cervical polyp (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Colpocele (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Epididymitis (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatic obstruction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 4 (4) | 1 (1)
Prostatomegaly (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Rectocele (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Testicular cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Uterine prolapse (Reproductive system and breast disorders) | 2 (2) | 1 (2)
Uterovaginal prolapse (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Acute lung injury (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 12 (12)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 15 (20)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Bullous lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 53 (79) | 71 (88)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 24 (24) | 18 (19)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 8 (9)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 0 (0)
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nocturnal dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Pharyngeal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 5 (5)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 10 (10)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 11 (11)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (5)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 8 (8)
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Reflux laryngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 11 (13) | 9 (10)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2)
Snoring (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 23 (25) | 22 (24)
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dry gangrene (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dyshidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Keloid scar (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Neurodermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Neuropathic ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Panniculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Scar pain (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin fibrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin necrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Skin reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 22 (24) | 21 (22)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Coronary revascularisation (Surgical and medical procedures) | 1 (1) | 2 (2)
Percutaneous coronary intervention (Surgical and medical procedures) | 1 (1) | 0 (0)
Accelerated hypertension (Vascular disorders) | 2 (2) | 0 (0)
Aortic aneurysm (Vascular disorders) | 8 (8) | 4 (4)
Aortic calcification (Vascular disorders) | 0 (0) | 1 (1)
Aortic occlusion (Vascular disorders) | 0 (0) | 2 (2)
Aortic stenosis (Vascular disorders) | 7 (7) | 4 (4)
Arterial insufficiency (Vascular disorders) | 1 (1) | 0 (0)
Arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 5 (5) | 2 (2)
Arteriovenous fistula (Vascular disorders) | 0 (0) | 1 (1)
Blood pressure inadequately controlled (Vascular disorders) | 1 (1) | 1 (1)
Circulatory collapse (Vascular disorders) | 1 (1) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 9 (9) | 8 (8)
Diabetic macroangiopathy (Vascular disorders) | 1 (1) | 0 (0)
Embolism venous (Vascular disorders) | 1 (1) | 0 (0)
Extremity necrosis (Vascular disorders) | 3 (3) | 6 (6)
Femoral artery embolism (Vascular disorders) | 1 (1) | 0 (0)
Femoral artery occlusion (Vascular disorders) | 7 (8) | 2 (2)
Granulomatosis with polyangiitis (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 3 (3) | 5 (5)
Haemorrhage (Vascular disorders) | 0 (0) | 3 (3)
Haemorrhagic infarction (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 30 (33) | 29 (32)
Hypertensive crisis (Vascular disorders) | 16 (17) | 17 (18)
Hypertensive emergency (Vascular disorders) | 3 (3) | 2 (2)
Hypoperfusion (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 17 (18) | 19 (22)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 3 (3)
Iliac artery occlusion (Vascular disorders) | 2 (2) | 1 (1)
Intermittent claudication (Vascular disorders) | 10 (11) | 10 (11)
Necrosis ischaemic (Vascular disorders) | 1 (2) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 5 (6) | 6 (6)
Peripheral arterial occlusive disease (Vascular disorders) | 43 (49) | 24 (25)
Peripheral artery aneurysm (Vascular disorders) | 3 (3) | 1 (1)
Peripheral artery dissection (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery stenosis (Vascular disorders) | 8 (9) | 18 (20)
Peripheral artery thrombosis (Vascular disorders) | 2 (2) | 2 (2)
Peripheral embolism (Vascular disorders) | 2 (2) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 39 (46) | 24 (35)
Peripheral vascular disorder (Vascular disorders) | 20 (22) | 21 (24)
Shock (Vascular disorders) | 0 (0) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 1 (1)
Subclavian artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Subclavian artery stenosis (Vascular disorders) | 2 (2) | 0 (0)
Thrombophlebitis (Vascular disorders) | 1 (1) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 3 (3)
Varicose vein (Vascular disorders) | 1 (1) | 2 (2)
Vascular occlusion (Vascular disorders) | 1 (1) | 0 (0)
Vascular stenosis (Vascular disorders) | 1 (1) | 1 (1)
Vasculitis (Vascular disorders) | 0 (0) | 1 (1)
Venous insufficiency (Vascular disorders) | 1 (1) | 1 (1)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=8212) | Saxagliptin (N=8280)
Anaemia (Blood and lymphatic system disorders) | 198 (208) | 197 (204)
Angina pectoris (Cardiac disorders) | 197 (217) | 171 (188)
Constipation (Gastrointestinal disorders) | 164 (175) | 170 (183)
Diarrhoea (Gastrointestinal disorders) | 314 (369) | 321 (379)
Nausea (Gastrointestinal disorders) | 182 (215) | 200 (218)
Fatigue (General disorders) | 192 (215) | 167 (179)
Oedema peripheral (General disorders) | 352 (375) | 343 (380)
Bronchitis (Infections and infestations) | 375 (453) | 331 (414)
Influenza (Infections and infestations) | 195 (232) | 199 (230)
Nasopharyngitis (Infections and infestations) | 280 (334) | 293 (341)
Upper respiratory tract infection (Infections and infestations) | 324 (398) | 330 (408)
Urinary tract infection (Infections and infestations) | 323 (431) | 307 (389)
Diabetes mellitus (Metabolism and nutrition disorders) | 666 (834) | 538 (666)
Hyperglycaemia (Metabolism and nutrition disorders) | 278 (327) | 215 (271)
Arthralgia (Musculoskeletal and connective tissue disorders) | 306 (332) | 313 (354)
Back pain (Musculoskeletal and connective tissue disorders) | 319 (350) | 330 (358)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 165 (179) | 168 (185)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 321 (342) | 264 (298)
Dizziness (Nervous system disorders) | 344 (393) | 374 (485)
Headache (Nervous system disorders) | 241 (255) | 208 (240)
Cough (Respiratory, thoracic and mediastinal disorders) | 302 (337) | 258 (282)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 199 (217) | 182 (196)
Hypertension (Vascular disorders) | 321 (352) | 349 (379)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AstraZeneca's Publication Policy, data disclosure and transparency are available at the website: http://www.astrazeneca.com/responsibility/code-and-policies/policies?itemId=4861823&nav=yes. All papers or abstracts must be submitted to the Steering Committee and the SPONSOR, through BRIGHAM, for review of its appropriateness and scientific merit at least six weeks prior to submission to any publication.